CLINICAL TRIAL: NCT05997758
Title: Investigating Surprise Signals in the Anterior Insula in Epilepsy Patients With Stereoelectroencephalography Recording
Brief Title: Investigating Surprise Signals in the Anterior Insula
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Fabienne PICARD, Prof, University Hospital, Geneva
Other Study IDs: 2022-02041
Record Dates: First submitted 2023-06-01; First posted 2023-08-18 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Drug Resistant Epilepsy; Healthy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients who suffer from potentially surgically remediable drug-resistant focal epilepsy and who require evaluation with intracranial stereo-EEG electrodes and have them implanted in the anterior insula.
  N = 10
  Interventions: Other: SEEG stimulation; Behavioral: Adaptation task
- Subclinical: Healthy individuals who match the clinical population in age and level of education.
  N = 40
  Interventions: Behavioral: Adaptation task

INTERVENTIONS:
Other: SEEG stimulation — Electrodes already implanted in patient's anterior insula will be stimulated below the patient-specific threshold at which a seizure was induced. This stimulations will coincide with certain trials in the adaptation task.
  Groups: Patients
Behavioral: Adaptation task — Participants will perform a task that requires them to learn and correctly respond to outliers of two sorts; inconsequential outliers, which require no action, and outliers that are relevant to the course of stimuli and outcomes in future trials, requiring adaptive action.

SUMMARY:
The investigators propose a behavioral experiment with SEEG recording and stimulation, to both confirm the role of a brain region known as the anterior insula in identifying surprise, and disambiguate between competing principles behind adaptation: optimizing and satisficing. Optimizers continue to learn and adapt if performance can be improved, while satisficers are satisfied with a good enough performance and will cease adapting once that is reached.

To study surprise signals in the anterior insula, a brain structure where these signals have been very prominent, the investigators will employ an experiment with subjects who are under SEEG (stereoelectroencephalogram) recording, that is, recording from electrodes which have been surgically implanted in the brain. These recordings will be done as patients perform a task where they try to anticipate the movements of a target on a line in two different learning environments (conditions). The experimenters will then determine whether these signals reflect surprise relative to past engagement with the environment, or surprise that reveals that the agent no longer feels in control because uncertainty is not in line with the reference model. If evidence is consistent with the former, adaptation reflects traditional reinforcement and aims at optimizing behavior. If evidence instead is consistent with the latter, behavior is guided by a prior model (a reference model) and behavior is satisficing.

An fMRI study by d'Acremont and Bossaerts provides initial evidence that activation in the anterior insula supports the satisficing hypothesis, however it lacks the temporal granularity to completely rule out optimizing. In the current project, the investigators propose to use the higher time resolution of SEEG recordings to confirm these findings and reject the optimizing hypothesis.

Additionally, stimulations of the anterior insula during a subset of trials will be used to determine whether insular activation following surprise signals and preceding changes in behavior (learning) is merely correlational or in fact causal. Stimulation will allow us to determine to what extent the subjects' sense of control and subsequent behavior can be influenced in accordance with surprise-based modeling of behavior.

The cohort for this study will be patients with drug-resistant, focal epilepsy and who are hospitalized at the Hôpitaux Universitaires de Genève (HUG) for pre-surgical evaluation of their epilepsy using SEEG. The protocol will run in parallel with the patients' clinical procedures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Fluent in French or English
* Patient who suffers from potentially surgically remediable drug-resistant focal epilepsy
* Patient who requires evaluation with intracranial stereo-EEG electrodes and has them implanted in the anterior insula
* Patient who is able and willing to provide informed consent

Exclusion Criteria:

* Severe concomitant psychiatric disease or major psychological distress
* Patients who have an implanted stimulation device (e.g. pacemaker, defibrillator, neurostimulator)
* Intellectual/neurological/psychiatric deficiencies* or inability to understand or follow the procedure
* Visual/motor deficiencies which could affect task performance
* The presence of seizures during routine clinical stimulation of insular electrodes
* Failure to complete the pre-experiment task training

  * As determined by their clinical evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who suffer from potentially surgically remediable drug-resistant focal epilepsy and require evaluation with intracranial stereo-EEG electrodes and have them implanted in the anterior insula hospitalized at the Hôpitaux Universitaires Genève.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Bias adjustment -- non-stimulation trials (behavioral, numerical) | Up to 2500 ms after stimuli presentation. All data collected during eight 5-minute sessions on the same day
  Subjects' choices, measured as the degree of bias correction they employ (a numerical value typically between 0 and +/-3) during outlier trials and the trials immediately following them. These will be quantitatively compared between conditions using Bayes-optimal choices and choices as predicted by Model-Reference Based Adaptive Control.
Bias adjustment -- stimulation trials (behavioral, numerical) | Up to 2500 ms after stimuli presentation. All data collected during four 5-minute sessions on the same day
  Subjects' choices, measured as the degree of bias correction they employ (a numerical value typically between 0 and +/-3) during stimulation trials (both outlier and non-outlier trials). These will be quantitatively compared to choices on the same trial types without stimulation.
SEEG-ERP--non-stimulation trials | Up to 2500 ms after stimuli presentation. Averaged over all trials for each task condition. All data collected during 8 5-minute sessions on the same day
  Event-related potentials (ERPs) extracted from subjects' stereoelectroencephalographies from intercranial electrodes implanted in the anterior insulae. ERPs will be averaged across the time series and t-statistics will be computed for effect of condition (outlier type).
SEEG-TF--non-stimulation trials | Up to 2500 ms after stimuli presentation. Averaged over all trials for each task condition. All data collected during 8 5-minute sessions on the same day
  The stereoelectroencephalographies from intercranial electrodes implanted in subjects' anterior insulae will be used for time frequency (TF) analyses. Time series components will be extracted for multiple frequencies and t-statistics of the effects of condition (outlier type) will be computed for each frequency.

SECONDARY OUTCOMES:
Reaction time (numerical) | Up to 2500 ms after stimuli presentation. All data collected during 8 5-minute sessions on the same day
  Comparison of subjects' response times to stimuli

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Neurologie, Dpt des Neurosciences cliniques HUG, Geneva, Switzerland

REFERENCES:
- [Background] d'Acremont M, Bossaerts P. Neural Mechanisms Behind Identification of Leptokurtic Noise and Adaptive Behavioral Response. Cereb Cortex. 2016 Apr;26(4):1818-1830. doi: 10.1093/cercor/bhw013. Epub 2016 Feb 4. PMID 26850528